CLINICAL TRIAL: NCT05897099
Title: Comprehensive HIV and Harm Prevention Via Telehealth: CHARIOT, a Randomized Controlled Trial
Brief Title: Comprehensive HIV and Harm Prevention Via Telehealth
Acronym: CHARIOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Hansel Tookes, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20230061; R01DA058352 (NIH)
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Tele-harm Reduction (Experimental): Participants will have enhanced access to a physician and clinical psychologist via remote video technology wherever the participant is located and prefers engagement (SSP, home, shelter, encampment). Participants will be in this group for 12 months.
  Interventions: Behavioral: Comprehensive Tele-harm Reduction
- Off-site Linkage to HIV prevention (Active Comparator): Participants in this group will receive off-site linkage to HIV care by having case management/social work services through our community engagement team. Participants will be in this group for 12 months.
  Interventions: Behavioral: Off-site Linkage to HIV Prevention

INTERVENTIONS:
Behavioral: Comprehensive Tele-harm Reduction — Comprehensive Tele-Harm Reduction is on-demand services including low-barrier access to PrEP, medications for substance use disorder and hepatitis C treatment. It includes mobile phlebotomy, peer harm reduction counseling, medication management, telehealth mental health/substance use disorder services-- all delivered via an syringe services program.
  Arms: Comprehensive Tele-harm Reduction
Behavioral: Off-site Linkage to HIV Prevention — The community engagement team is comprised of peers and social workers and provides the wraparound support needed.The team will assist participants in scheduling appointments at community health clinics. The community engagement team provides active clinic referral- that is, a member of the team will accompany patients to the first clinic visit.
  Arms: Off-site Linkage to HIV prevention

SUMMARY:
The purpose of this study is to test 2 different ways to offer medications to prevent human immunodeficiency virus (HIV), cure hepatitis C virus (HCV) (if applicable) and treat substance use disorder (if desired) in people who inject drugs.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* able to speak English or Spanish
* willing and able to sign informed consent, provide locator information and medical records release
* non-reactive result on rapid HIV test
* use of SSP to exchange syringes 2 times in the past 3 months
* planning to stay in the area for 12 months

Exclusion Criteria:

* reactive HIV test
* currently on medications for opioid use disorder (MOUD) by urine drug screen
* currently on PrEP by self-report
* Principal or site investigator discretion
* currently in prison or jail
* current enrollment in Clinical Trials Network 121
* receipt of tele-harm reduction in previous 3 months
* signs or symptoms of acute HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
HIV prevention via pre-exposure prophylaxis (PrEP) | up to 12 months
  Intracellular levels of tenofovir diphosphate (TFV-DP) by DBS or cabotegravir injection in previous 8 weeks or lenacapavir injection in previous 6 months by electronic health record abstraction
HIV prevention via medications for opioid use disorder | up to 12 months
  Buprenorphine/norbuprenorphine or methadone on urine drug screen; or naltrexone or buprenorphine extended-release injection in previous 4 weeks by electronic health record abstraction

SECONDARY OUTCOMES:
syringe coverage | up to 12 months
  Number of syringes distributed/(number of injections per day x days between exchanges)
PrEP Adherence | up to 12 months
  TFV-DP level of 700 fmol/punch on DBS for Truvada; TFV-DP level of 950 fmol/punch on DBS for Descovy
Engagement in HCV treatment | Up to 12 months
  Direct acting antiviral prescription confirmed on electronic health record abstraction
HCV cure | up to 12 months
  Negative HCV RNA viral load at least 12 weeks post treatment completion
treatment of sexually transmitted infections | up to 12 months
  Medical records show prescription of appropriate antibiotics
time to harm | up to 12 months
  Time to: (1) emergency department visit or hospitalization for injection-related infection or overdose; (2) incident HIV infection; (3) incident HCV infection; or (4) death from overdose
number of harms | up to 12 months
  Count of (1) emergency department visit or hospitalization for injection-related infection or overdose; (2) incident HIV infection; (3) incident HCV infection; or (4) death from overdose

CONTACTS AND LOCATIONS:
Overall Officials: Hansel Tookes, MD, Principal Investigator — University of Miami; Tyler Bartholomew, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - IDEA Miami, Miami, Florida
  - IDEA Syringe Services Program, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartholomew TS, Plesons M, Serota DP, Alonso E, Metsch LR, Feaster DJ, Ucha J, Suarez E Jr, Forrest DW, Chueng TA, Ciraldo K, Brooks J, Smith JD, Barocas JA, Tookes HE. Project CHARIOT: study protocol for a hybrid type 1 effectiveness-implementation study of comprehensive tele-harm reduction for engagement of people who inject drugs in HIV prevention services. Addict Sci Clin Pract. 2024 Mar 25;19(1):21. doi: 10.1186/s13722-024-00447-9. PMID 38528570